CLINICAL TRIAL: NCT01700894
Title: Reducing Health Disparities in African American Women: Lifestyle Physical Activity Adherence
Brief Title: Women's Walking Program
Acronym: WWP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, JoEllen Wilbur, PhD, APN, FAAN, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09021301-IRB01; R01NR004134 (NIH)
Record Dates: First submitted 2012-09-28; First posted 2012-10-04 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Cardiovascular Diseases
Keywords: Physical Activity; African American; Adherence
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Walking Program + motivational interviewing calls (Experimental): The Women's Walking Program (WWP) core included a lifestyle PA prescription with an accelerometer for self-feedback and monitoring and 6 group visits (1 every week for 5 weeks in the 1st 24 weeks and 1 3 months later) targeted to increase lifestyle PA in AA women.
  Participant in the WWP plus motivational interviewing telephone call arm receives 11 motivational interviewing telephone calls from an interventionist, with two calls in between each of the group-visits. Motivational interviewing calls are tailored to the individual and intended to sustain intervention effects between group-visits
  Interventions: Behavioral: Walking Program + Motivational Interviewing Calls
- Walking Program + automated calls (Experimental): The Women's Walking Program (WWP) core, including a lifestyle physical activity prescription with an accelerometer for self-feedback and monitoring and 6 group visits (1 every 5 weeks during the first 24 weeks and 1 3 months later) targeted to increase lifestyle physical activity in African American women.
  Participants in the WWP plus automated telephone call arm receive 11 automated calls with two calls sent between each group-visit. The automated calls are intended to supplement and sustain the intervention effects of the group-visits.
  Interventions: Behavioral: Walking Program + Automated Calls
- Walking Program (Experimental): The Women's Walking Program (WWP) core, including a lifestyle physical activity prescription with an accelerometer for self-feedback and monitoring and 6 group visits (1 every 5 weeks during the first 24 weeks and 1 3 months later) targeted to increase lifestyle physical activity in African American women.
  Participants in the WWP receive no telephone calls.
  Interventions: Behavioral: Walking Program

INTERVENTIONS:
Behavioral: Walking Program + Motivational Interviewing Calls
  Arms: Walking Program + motivational interviewing calls
Behavioral: Walking Program + Automated Calls
  Arms: Walking Program + automated calls
Behavioral: Walking Program
  Arms: Walking Program

SUMMARY:
African American (AA) women have the lowest physical activity (PA) levels, which contributes to substantial disparities in cardiovascular health and depressive symptoms. There is a need to examine ways to promote PA that are appealing, applicable to clinical practice, and cost-effective. The purpose of this clinical trial is to test the efficacy of the Women's Walking Program (WWP), consisting of a lifestyle PA prescription and "group visit" delivery model, with or without tailored telephone contacts between group visits for increasing adherence to PA and improving health outcomes. Two telephone contact strategies will be compared against a no-telephone control condition: a person-administered contact strategy using brief motivational interviewing and an automated contact strategy using a telephone computer-linked system. Group visits and telephone contacts are designed to increase adherence to lifestyle PA with an emphasis on accumulation of 3,000 steps daily over baseline. The aims of this study are (1) to compare the initial (adoption 24 weeks) and longer-term (maintenance 2nd 24 weeks) effectiveness of the WWP plus person-administered telephone contacts, WWP plus automated telephone contacts, and the WWP without telephone contacts on (a) increasing adherence to lifestyle PA, (b) improving health outcomes (aerobic fitness, body composition, depressive symptoms), (c) improving self-efficacy (confidence in one's ability to be physically active) and outcome expectations (expected benefits to being more active); and (2) to compare cost-effectiveness of the three telephone treatment conditions in relation to adherence to lifestyle PA and health outcomes.

The investigators will randomly assignment of the order of administering the three conditions to six community health care sites. These six sites are similar with respect to race, socioeconomic status, and residential mobility. The study will include 288 sedentary AA women aged 40 to 65 years who have no major signs or symptoms of cardiovascular disease (CVD); no history of myocardial infarction, stroke, or diabetics with elevated HgA1c; BP < 160/100.

Initial screening will occur in person or over the phone. Further screening at the data collection site with an advanced practice nurse will include blood work for glucose and lipoproteins, a history and physical, and resting EKG. At baseline, 24 and 48 weeks all women who are eligible will: be given questionnaires on physical activity, health and factors that influence their physical activity; have their height, weight, waist circumference measured; and do a two minute step test. All three treatment group will attend 5 group visits every 5 weeks during adoption (first 24 weeks) and 1 booster group visit during maintenance (week 36). The group visit consists of brief individual time with a staff member followed by a group visit with motivational videotapes. All treatment groups will self-monitor their physical activity with accelerometers and enter their step data into a voice response system.

The groups receiving the automated telephone contact strategy and the group receiving the person telephone contact strategy will have the same number and spacing of the telephone contacts (nine 10- to 15-minute telephone contacts delivered every two to three weeks between group visits during adoption and two telephone contacts [weeks 28, 43] during maintenance). Using motivational interviewing, a nurse will tailor the telephone discussion to the person telephone contact group to match the participant's needs, experiences, barriers, motivation, and confidence. Women in the automated telephone contact group will receive an automated call with feedback on their progress based on the information they reported into the ATCL system. The automated telephone contact system will deliver feedback on progress, problem solving, goal-setting, and support. All information will be delivered in the voice of one of our staff members. The third treatment group will receive no telephone contacts between group visits.

Potential risks exist for women who have medical problems, which contraindicate physical exercise. Additional risks associated with the walking program include safety and injury. There are potential risks of infection at the site of the one time finger blood withdrawal. Potential benefits to subjects include improved aerobic fitness, blood cholesterol, body composition and blood pressure and fewer symptoms. The subjects will be given a physical activity prescription that should benefit them through life and decrease their risk for CVD.

Women will be recruited throughout the West and South side of Chicago. They will give verbal consent at the screening questionnaire and sign an informed consent at the time of the screening history and physical. They will be told that participation is voluntary, they may decline or withdraw at will at any time, and all results will be held strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* AA female
* sedentary: Sedentary will be defined as no participation in regular planned (3 or more times a week) moderate (e.g., walking) or vigorous (e.g., jogging, speed walking) in the past 6 months.
* aged 40 to 65 years
* able to commit to attending the study group visits and have a telephone
* without disabilities that would prevent regular participation in PA such as walking as determined by the PARQ and baseline screening. PA

Exclusion Criteria:

* Women will be excluded from the study if they have major signs or symptoms of CV disease
* a history of myocardial infarction, stroke or Type 1 diabetes
* BP >160/100
* HgA1 >9 ( done on diabetics only)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Adherence to physical activity prescription | baseline, 24, and 48 weeks
  The investigators will compare the effects at 24 weeks and 48 weeks of the WWP plus three telephone conditions on increasing adherence to lifestyle physical activity over baseline physical activity.

SECONDARY OUTCOMES:
Body Composition | 24 and 48 weeks from baseline
  The investigators will compare the effects at 24 weeks and 48 weeks of the WWP plus three telephone conditions on decreasing body composition over baseline body composition.
  Body Composition measured with body mass index
Depression | 24 and 48 weeks from baseline
  The investigators will compare the effects at 24 weeks and 48 weeks of the WWP plus three telephone conditions on improving depressive symptoms over baseline symptoms.
  Depression is measured with the CES-D.
Stress | 24 and 48 weeks from baseline
  The investigators will compare the effects at 24 weeks and 48 weeks of the WWP plus three telephone conditions on improving stress over baseline stress.
  Stress is measured with Cohen's measure of Global Perceived Stress.

CONTACTS AND LOCATIONS:
Overall Officials: JoEllen Wilbur, PhD, Principal Investigator — Rush University College of Nursing
Locations (7):
- United States (7):
  - University of Illinois at Chicago Mile Square Health Center at Back of the Yards, Chicago, Illinois
  - University of Illinois at Chicago Mile Square Health Center, Chicago, Illinois
  - Roseland Community Hospital, Chicago, Illinois
  - Holy Cross Hospital, Chicago, Illinois
  - Austin Health Center of Cook County Health & Hospitals System, Chicago, Illinois
  - Westside Health Authority, Chicago, Illinois
  - Rush Oak Park Hospital, Oak Park, Illinois

REFERENCES:
- [Derived] Garland M, Wilbur J, Fogg L, Halloway S, Braun L, Miller A. Self-Efficacy, Outcome Expectations, Group Social Support, and Adherence to Physical Activity in African American Women. Nurs Res. 2021 Jul-Aug 01;70(4):239-247. doi: 10.1097/NNR.0000000000000516. PMID 33870956
- [Derived] Wilbur J, Schoeny ME, Buchholz SW, Fogg L, Miller AM, Braun LT, Halloway S, Dancy BL. Women's Lifestyle Physical Activity Program for African American Women: Fidelity Plan and Outcomes. J Phys Act Health. 2016 Oct;13(10):1100-1109. doi: 10.1123/jpah.2015-0701. Epub 2016 Aug 16. PMID 27256816